CLINICAL TRIAL: NCT05435651
Title: A Randomized Clinical Trial to Assess The Effectiveness and Safety of Digital Therapy for Treating Attention Deficit Hyperactivity Disorder in Children
Brief Title: Digital Therapy for Treating Attention Deficit Hyperactivity Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SZLFADHD2022
Record Dates: First submitted 2022-06-23; First posted 2022-06-28 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Digital therapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: The present study will be carried out using a parallel randomized study design. Each participant will be randomly assigned either to Multitask game-based digital therapy or to Schulte Grid digital game control group.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multitask game-based digital therapy (Experimental): Multitask game-based digital therapy group will be asked to practice multitask-game on the system for approximately 25 minutes/day at least 5 days a week. Compliance will be monitored electronically.
  Interventions: Behavioral: Multitask game-based digital therapy
- Schulte Grid digital game (Active Comparator): Schulte Grid digital game group will be asked to practice Schulte Grid digital game on the system for approximately 25 minutes/day at least 5 days a week. Compliance will be monitored electronically.
  Interventions: Behavioral: Schulte Grid digital game

INTERVENTIONS:
Behavioral: Multitask game-based digital therapy — To practice multitask-game on the system for approximately 25 minutes/day at least 5 days a week.
  Arms: Multitask game-based digital therapy
Behavioral: Schulte Grid digital game — To practice Schulte Grid digital game on the system for approximately 25 minutes/day at least 5 days a week.
  Arms: Schulte Grid digital game

SUMMARY:
This study is designed to explore the effect of Multitask game-based digital therapy versus Schulte Grid digital game on attentional functioning (measured by the TOVA), ADHD symptoms, executive functioning, and clinical impairment, in children diagnosed with ADHD. Investigators will also evaluate the safety of digital therapy for intervention treatment of childhood attention deficit hyperactivity disorder.

DETAILED DESCRIPTION:
ADHD is a common neurodevelopmental disorder characterized by a persistent pattern of inattention and/or hyperactivity and impulsivity, resulting in functional impairment in multiple settings.The prevalence in China is estimated to be 6.26%. Front-line intervention for ADHD includes pharmacological and non-pharmacological interventions, which have shown short-term efficacy.There are limitations to current best practices for the treatment of ADHD.

Relating to pharmacotherapy, they are accompanied by adverse events in many children, do not normalize functioning , and adherence rates over time are generally low. Pharmacotherapy may not be suitable for some patients.Relating to non-pharmacological interventions, barriers to access limit the use of non-pharmacological interventions, given a shortage of properly trained paediatric mental health specialists and variability in insurance coverage for such services.

Digital therapy for ADHD may address these limitations with improved access, minimal side-effects, and low potential for abuse.There are studies show that digital intervention can significantly increase attentional functioning of children with ADHD.At present, there are few related researches on digital therapy in China.The total number of ADHD children is large in China, and electronic products are very popular in Chinese families.If digital therapies suitable for ADHD children in China can be developed, it will be of great significance for the promotion of human health.

Therefore, investigators designed the study to explore the effect of Multitask game-based digital therapy versus Schulte Grid digital game on attentional functioning (measured by the TOVA), ADHD symptoms, executive functioning, and clinical impairment, in children diagnosed with ADHD in China.Safety, tolerability, and compliance were also assessed.

The study will be a blinded (investigators and outcome assessors), randomized, parallel group, follow-up study of the sustained effects of 28 days of treatment with either Multitask game-based digital therapy or Schulte Grid digital game.

The trial will consist of 3 visits: Screening, FU-Day 14 visit and FU-Day 28 visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 years to 12 years, inclusive, at the time of parental informed consent.
* Male or female.
* Confirmed ADHD diagnosis , any presentation , at Screening based on DSM-V criteria and established via the MINI-KID administered by a trained clinician.
* Screening/Baseline score on the clinician-rated ADHDRS-IV score 24.
* Screening/Baseline score on the TOVA API -1.8.
* Not undergoing pharmacological treatment with methylphenidate or amphetamine-based products at time of Screening ; or, if undergoing pharmacolog ical treatment , must be willing and appropriate (i.e. not optimally treated in the investigator's judgment) to wash out of current regimen.
* Estimated IQ score~ 80 as assessed by Wechsler Intelligence Scale for Children-Fourth Edition ,WISC-IV.
* Ability to comply with all the testing and requirements.

Exclusion Criteria:

* Current, controlled (requiring a restricted medicatio n) or uncontrolled, comorbid psychiatric diagnosis , based on MINI-KID and subsequent clinical interviewing, with significant symptoms including but not limited to post-traumatic stress disorder , psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder , conduct disorder , or other symptomatic manifestatio ns that in the opinion of the Investigator may confound study data/assessments .
* Children who are currently at risk of suicide or have attempted suicide; children who have a history of suicide or are currently exhibiting active suicidal ideation or self-harm.
* Unable to stop taking ADHD medication.
* Motor condition (e.g., physical deformity of the hands/arms ; prostheses) that prevents playing the digital therapy as reported by the parent or observed by the investigator .
* Recent history (within the past 6 months) of suspected substance abuse or dependence.
* History of seizures (exclusive of febr ile seizures) , or significant motor or vocal tics, including but not limited to Tourette 's Disorder.
* Diagnosis of or parent-reported color blindness.
* Uncorrected visual acuity (Confirmed in-clinic via ability of subject to play the game).
* With severe mental retardation.
* Any other medical condition that in the opinion of the investigato r may confound study data/assessments.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-07-16 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
the TOVA API | Baseline
  The primary outcome measure was the mean change in The Attention Performance Index (API) of TOVA. The TOVA is a validated, computerised, continuous performance test that objectively measures attention and inhibitory control, normalised by age and sex.
  The API is calculated from variability, response time, and d' (D Prime) using the following formula: API = Response Time Z score (Half 1) + d' Z score (Half 2) + Variability Z score (Total) + 1.80
  API tells how similar the score is to the ADHD profile. A score of less than 0 indicates that the subject had similar performance to a normative ADHD population. A lower score indicates a more severe ADHD profile.
the TOVA API | 14 days after enrollment
  The primary outcome measure was the mean change in The Attention Performance Index (API) of TOVA. The TOVA is a validated, computerised, continuous performance test that objectively measures attention and inhibitory control, normalised by age and sex.
  The API is calculated from variability, response time, and d' (D Prime) using the following formula: API = Response Time Z score (Half 1) + d' Z score (Half 2) + Variability Z score (Total) + 1.80
  API tells how similar the score is to the ADHD profile. A score of less than 0 indicates that the subject had similar performance to a normative ADHD population. A lower score indicates a more severe ADHD profile.
the TOVA API | 28 days after enrollment
  The primary outcome measure was the mean change in The Attention Performance Index (API) of TOVA. The TOVA is a validated, computerised, continuous performance test that objectively measures attention and inhibitory control, normalised by age and sex.
  The API is calculated from variability, response time, and d' (D Prime) using the following formula: API = Response Time Z score (Half 1) + d' Z score (Half 2) + Variability Z score (Total) + 1.80
  API tells how similar the score is to the ADHD profile. A score of less than 0 indicates that the subject had similar performance to a normative ADHD population. A lower score indicates a more severe ADHD profile.

SECONDARY OUTCOMES:
The ADHD-Rating Scale | Baseline
  The ADHD-Rating Scale is an 18-item scale assessing the frequency of each ADHD symptom based on DSM-IV criteria. The scale consists of 2 subscales: inattention (9 items) and hyperactivity-impulsivity (9 items). Each item is scored on a 4-point scale ranging from 0 (rarely or never) to 3 (very often) with total scores ranging from 0-54. A higher score indicates more severe ADHD symptoms and behaviors.
The ADHD-Rating Scale | 14 days after enrollment
  The ADHD-Rating Scale is an 18-item scale assessing the frequency of each ADHD symptom based on DSM-IV criteria. The scale consists of 2 subscales: inattention (9 items) and hyperactivity-impulsivity (9 items). Each item is scored on a 4-point scale ranging from 0 (rarely or never) to 3 (very often) with total scores ranging from 0-54. A higher score indicates more severe ADHD symptoms and behaviors.
The ADHD-Rating Scale | 28 days after enrollment
  The ADHD-Rating Scale is an 18-item scale assessing the frequency of each ADHD symptom based on DSM-IV criteria. The scale consists of 2 subscales: inattention (9 items) and hyperactivity-impulsivity (9 items). Each item is scored on a 4-point scale ranging from 0 (rarely or never) to 3 (very often) with total scores ranging from 0-54. A higher score indicates more severe ADHD symptoms and behaviors.
The Clinical Global Impression Scale - Improvement (CGI-I) | 14 days after enrollment
  The Clinical Global Impression Scale - Improvement (CGI-I) is a clinician's comparison of the participant's overall clinical condition at follow up to the overall clinical condition at baseline. The CGI-S is a 7-point scale where 1 = Very much improved, 2=Much improved, 3=Minimally improved, 4=No change, 5=Minimally worse, 6=Much worse, and 7=Very much worse.
  A score of 1, 2, or 3 would indicate overall improvement of ADHD severity.
The Clinical Global Impression Scale - Improvement (CGI-I) | 28 days after enrollment
  The Clinical Global Impression Scale - Improvement (CGI-I) is a clinician's comparison of the participant's overall clinical condition at follow up to the overall clinical condition at baseline. The CGI-S is a 7-point scale where 1 = Very much improved, 2=Much improved, 3=Minimally improved, 4=No change, 5=Minimally worse, 6=Much worse, and 7=Very much worse.
  A score of 1, 2, or 3 would indicate overall improvement of ADHD severity.
BRIEF Inhibit Percentile | Baseline
  The Behavior Rating Inventory of Executive Function (BRIEF) is a parent-rated form that assesses everyday behavior associated with specific domains of the executive functions of their child. The BRIEF working memory metacognition subscale measures the participants ability to hold information when completing a task in a sequential manner.
  A lower subscale score indicates better ability of working memory.
BRIEF Inhibit Percentile | 14 days after enrollment
  The Behavior Rating Inventory of Executive Function (BRIEF) is a parent-rated form that assesses everyday behavior associated with specific domains of the executive functions of their child. The BRIEF working memory metacognition subscale measures the participants ability to hold information when completing a task in a sequential manner.
  A lower subscale score indicates better ability of working memory.
BRIEF Inhibit Percentile | 28 days after enrollment
  The Behavior Rating Inventory of Executive Function (BRIEF) is a parent-rated form that assesses everyday behavior associated with specific domains of the executive functions of their child. The BRIEF working memory metacognition subscale measures the participants ability to hold information when completing a task in a sequential manner.
  A lower subscale score indicates better ability of working memory.
Adverse Device Effects | 14 days after enrollment
  The expectedness of an ADE shall be documented in case Report Form（CRF）. 1. Dizziness,2. Nausea,3. Headache,4. Increased and unusual levels of frustration during game play.
Adverse Device Effects | 28 days after enrollment
  The expectedness of an ADE shall be documented in case Report Form（CRF）. 1. Dizziness,2. Nausea,3. Headache,4. Increased and unusual levels of frustration during game play.

CONTACTS AND LOCATIONS:
Overall Officials: Daqian Zhu, PhD, Study Chair — Department of Psychological Medicine, Children's Hospital of Fudan University
Locations (1):
- Children's hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kollins SH, DeLoss DJ, Canadas E, Lutz J, Findling RL, Keefe RSE, Epstein JN, Cutler AJ, Faraone SV. A novel digital intervention for actively reducing severity of paediatric ADHD (STARS-ADHD): a randomised controlled trial. Lancet Digit Health. 2020 Apr;2(4):e168-e178. doi: 10.1016/S2589-7500(20)30017-0. Epub 2020 Feb 24. PMID 33334505
- [Background] Kollins SH, Childress A, Heusser AC, Lutz J. Effectiveness of a digital therapeutic as adjunct to treatment with medication in pediatric ADHD. NPJ Digit Med. 2021 Mar 26;4(1):58. doi: 10.1038/s41746-021-00429-0. PMID 33772095
- [Background] Davis NO, Bower J, Kollins SH. Proof-of-concept study of an at-home, engaging, digital intervention for pediatric ADHD. PLoS One. 2018 Jan 11;13(1):e0189749. doi: 10.1371/journal.pone.0189749. eCollection 2018. PMID 29324745